CLINICAL TRIAL: NCT00471315
Title: Pilot Study of the Efficacy and Tolerability of Duloxetine in Patients With Suspected Functional Pancreatic/Biliary Pain (Sphincter of Oddi Dysfunction).
Brief Title: Duloxetine in Patients With Suspected Functional Pancreatic/Biliary Pain (Sphincter of Oddi Dysfunction)
Acronym: SOD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR16489
Record Dates: First submitted 2007-05-08; First posted 2007-05-09 (Estimated); Results first posted 2014-02-06 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Sphincter of Oddi Dysfunction
Keywords: SOD; Common Bile Duct Diseases; Sphincterotomy; Cholangiopancreatography, Endoscopic Retrograde
MeSH Terms: conditions — Sphincter of Oddi Dysfunction; Common Bile Duct Diseases | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Duloxetine (No Intervention): A preliminary, open-label single center study of duloxetine in patients with SOD
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — A preliminary, open-label single center study of duloxetine in patients with SOD
  Other Names: Cymbalta

SUMMARY:
Open-label single center study of duloxetine in patients with SOD who have failed to respond to the standard treatments.

This protocol is designed to explore the tolerability and efficacy of Duloxetine in the management of patients with known or suspected Sphincter of Oddi dysfunction (SOD).

DETAILED DESCRIPTION:
SOD is a disorder involving the bile duct or pancreas causing a burning pain or cramping in the epigastric (upper stomach) area that can radiate (spread) to the back or under the right shoulder blade. This discomfort is thought to be caused by tightening of the Sphincter of Oddi, which is the muscle opening that controls the flow of bile and juices from the pancreas (enzymes) into the small intestine. It can also be caused by contractions of the common bile duct (the duct that allows bile from the liver into the small intestine).

The purpose of this research is to study how well a medication called Duloxetine works when used to treat pain associated with SOD. Duloxetine (also called Cymbalta) is a medication approved by the FDA for the treatment of depression and for the treatment of pain caused by nerve damage associated with diabetes. However, for the purposes of this research, Duloxetine is considered investigational (experimental) since it will test how well this medication works for the treatment of pain associated with SOD. (Cymbalta replaced with Duloxetine in remainder of consent as requested).

PRIMARY OBJECTIVE

● Treatment effect as measured by the global assessment of change (PGIC) after 3 months of treatment with duloxetine.

SECONDARY OBJECTIVES

* Toleration of the medication as measured by the duloxetine compliance rate;
* Safety as recorded by adverse events (AEs)
* Effect of treatment on pain reduction as measured by a pain burden assessment tool (RAPID 3 & RAPID 1-Month);
* Effect of treatment on quality of life (QOL) as measured by the SF-36.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients referred to MUSC pancreatico-biliary service for investigation/ mgt of functional upper abdominal pain symptoms;
* No clinically significant medical condition(s) as determined by the investigator;
* Symptom severity. At least 2 pain attacks in the previous month, with severity of at least 4/10 on the RAPID Start scale;
* Prior cholecystectomy;
* Age 18-65*;
* Functional pain characteristics as defined by Rome III Criteria;
* Structural causes of pain excluded by standard imaging and laboratory investigations;
* No clinically significant ECG results as determined by the investigator;
* All patients will give verbal and written Informed consent;
* Female patients must use an acceptable form of contraception, or be 2 years postmenopausal or surgically sterile*; and
* Geographically accessible for follow-up visits

EXCLUSION CRITERIA:

* History of/current psychosis, bipolar disorder, suicidal ideation or judged to be a significant suicide risk, as determined via baseline psychiatric assessment utilizing the MINI interview
* History of alcohol or any psychoactive substance abuse or dependence within the past 6 months, as determined via baseline psychiatric assessment utilizing the MINI interview
* Abnormal Liver Function Tests (> 3 x ULN)
* Known hypersensitivity to Duloxetine or any of the inactive ingredients
* Treatment with a monoamine oxidase inhibitor (MAOI) within 14 days of randomization or potential need to use an MAOI during study or within 5 days of discontinuation of study drug
* Treatment with fluoxetine (deleted MAOI) within 30 days of medication start date
* Treatment with excluded medications within 7 days prior to study medication start-up date
* Serious medical illness, including any cardiovascular, hepatic, renal respiratory hematologic, endocrinologic or neurologic disease, or significant laboratory abnormality as judged by study physician/investigator.
* Uncontrolled narrow-angle glaucoma
* Acute liver injury (such as hepatitis) or severe cirrhosis
* Prior lack of tolerability to duloxetine
* Pregnancy and breastfeeding

Participation in the study is approximately 4 months. There are 4 clinic visits and 2 telephone visits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Lawrence, MD, Principal Investigator — MUSC Digestive Disease Center
Locations (1):
- Digestive Disease Center, Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- See also: MUSC Digestive Disease Center Website — http://www.ddc.musc.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Duloxetine: Duloxetine orally in a dose of 30 mg/day in AM for the first week and 60 mg/day in AM thereafter.
Period: Overall Study
Arm/Group | Duloxetine
Started | 18
Completed | 10
Not Completed | 8
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Duloxetine
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Secondary Outcome: Toleration of the Medication as Measured by the Duloxetine Compliance Rate
Description: The secondary outcome measure of the study was number of patients who remained on Duloxetine at the completion of the study.
Time Frame: 3 Months
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 18
participants | 10

2. Primary Outcome: The Primary Outcome Measure Was a Patient Global Assessment of Change (PGIC) Scale.
Description: The primary outcome measure was a Patient Global Assessment of Change (PGIC) scale which reports the patient's overall view of any changes in their overall status since their sphincterotomy treatment. (1=Very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse). Success was defined as 3-month PGIC score of much or very much improved (PGIC of either 1 or 2). Patients missing the 3 month visit were considered failures for the primary outcome.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine
Number analyzed (Participants) | 18
units on a scale | 3.3 (1.32)

ADVERSE EVENTS:
Arm/Group | Duloxetine
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 11/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=18)
Fatigue (General disorders) | 11 (11)
Nausea (General disorders) | 10 (10)
Headaches (General disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 4 (4)
Decreased appetite (Gastrointestinal disorders) | 4 (4)
Insomnia (General disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
Most frequently reported adverse events included fatigue, nausea, headaches, constipation, decreased appetite and insomnia at primarily mild to moderate severity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No